CLINICAL TRIAL: NCT00081536
Title: A Phase I/II Study of Aroplatin and Capecitabine in Subjects With Unresectable Local Recurrence or Distant Metastases of Colorectal Cancer Refractory to 5-FU/Leucovorin and Irinotecan
Brief Title: Aroplatin and Capecitabine in Patients With Advanced Colorectal Cancer Resistant to Standard Therapies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aronex Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C-726-03
Record Dates: First submitted 2004-04-15; First posted 2004-04-20 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-04

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal Neoplasms; Colorectal Cancer; Colorectal Carcinoma; Colorectal Tumor; Neoplasms, Colorectal; Unresectable; Metastatic; Refractory
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — bis-neodecanoato-1,2-diaminocyclohexaneplatinum(II); Capecitabine

INTERVENTIONS:
Drug: Aroplatin (Liposomal NDDP) in combination with capecitabine

SUMMARY:
This study is a Phase I/II study. In Phase I of this study, the objective is to determine the maximum tolerated dose (MTD) of combination therapy with Aroplatin and capecitabine in subjects with unresectable, local recurrence or distant metastases of colorectal cancer refractory to 5-FU/leucovorin and irinotecan. In Phase II, the primary objective is to evaluate the response proportion and duration with Aroplatin/capecitabine therapy. Secondary objectives are to evaluate frequency and severity of adverse events.

DETAILED DESCRIPTION:
Phase I Primary Objective:

* Determine the MTD of Aroplatin/capecitabine subjects with unresectable local recurrence or distant metastases of colorectal cancer refractory to 5-FU/LV and irinotecan.

Phase II Primary Objective:

* Evaluate the response proportion and duration with Aroplatin/capecitabine therapy.

Phase II Secondary Objective:

* Evaluate the frequency of adverse events.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed colorectal cancer: unresectable local recurrence or distant metastases;
* Measurable disease (RECIST criteria);
* Refractory to 5-FU / leucovorin and irinotecan as described below;
* No prior therapy with oxaliplatin, any other platinum or capecitabine;
* ECOG score 0-2 (Karnofsky 100-70%);
* Life expectancy of greater then or equal to 5 months;
* Adequate hematopoietic, liver and renal function;
* Women of child-bearing potential have to practice adequate contraception;
* Signed written informed consent;
* Subjects must be willing to be followed during the course of treatment/observation and follow-up.

Refractory metastatic colorectal cancer

The following subjects are regarded refractory to treatment:

* Those with progression while receiving 5-FU/LV/irinotecan;
* Those with progression on irinotecan after prior 5-FU/LV treatment;
* Progression within six months of adjuvant 5-FU/LV/irinotecan;
* Progression within six months of adjuvant 5-FU/LV followed by progression on irinotecan

Subjects must have received at least one or more commonly used 5-FU/leucovorin and irinotecan regimens. Prior adjuvant therapy is allowed including 5-FU/leucovorin or other fluoropyrimidines except capecitabine and irinotecan.

Exclusion criteria:

* Previously diagnosed brain metastases if symptomatic and requiring active therapy;
* Other cancers within the last five years, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri or basal or squamous cell carcinoma of the skin;
* Concurrent chemotherapy or immunotherapy;
* Prior therapy for colorectal cancer within one month of admission to the present study;
* Primary or secondary immunodeficiency or use of corticosteroids or other immunosuppressive medication;
* Any serious concomitant medical or mental illness requiring intense therapy and interfering with participation in this study;
* Women must not be pregnant or breast-feeding;
* No participation in any clinical trial involving investigational drugs within 1 month from enrollment into the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105